

# STATISTICAL ANALYSIS PLAN

# A Multicenter, Randomized, Double-Blind, Controlled Study of EXPAREL for Postsurgical Pain Management in Subjects Undergoing Open Lumbar Spinal Fusion Surgery

**Protocol No.:** 402-C-409

**IND No.:** 69,198

**Study Phase:** 4

**Study Drug:** EXPAREL (bupivacaine liposome injectable

suspension)

**Date/Version:** 2 August 2017 (Amendment 2)

Prepared by: Napoleon Oleka, PhD

Pharma Data Associates, LLC

**Sponsor:** Pacira Pharmaceuticals, Inc.

5 Sylvan Way

Parsippany, NJ 07054 Tel: 973-254-3560

#### Confidentiality Statement

The information contained in this document is confidential and the property of Pacira Pharmaceuticals, Inc. It should not be reproduced, revealed, or sent to third parties other than Institutional Review Boards/Independent Ethics Committees and the Investigator's research support staff participating in the conduct of the study without the prior written authorization of Pacira Pharmaceuticals, Inc.

# 1. SIGNATURE PAGE

| Napoleon Oleka, PhD Associate Director, Biostatistics Pharma Data Associates, LLC | 08MAR2018<br>Date |
|---|---|
| Cher Mp | 08 March 2018 |
| Chao Wang, PhD President and Principal Statistician Pharma Data Associates. LLC | Date |
| Vincent Yu, PhD Senior Director, Biometrics Pacira Pharmaceuticals, Inc. | Date |
| 22 | 3/15/18 |
| Simon Dagenais, MD PhD<br>Senior Medical Director, Clinical Research | Date |
| Richard Scranton Picture Scranton Digitally signed by Richard Scranton DN: cn-Richard Scranton, o-Pacira No. cuchief Scientific Officer, enall-Richard-Scranton@pacira.com, c-US Date: 2216.03.16.075.31.31-04.007 | 3/16/2018 |
| Rich Scranton, MD, MPH<br>Chief Scientific Officer | Date |
| Michael Rozycki Digitally signed by Michael Rozycki DN: cn=Michael Rozycki, o=Regulatory Affairs, ou=Clinical Regulatory, email=michael.rozycki@pacira.com, c=US Date: 2018.03.1511:37:47-04'00' | |
| Michael Rozycki, PhD<br>Vice President, Regulatory Affairs and Pharmacovigil | Date<br>ance |

| 2. | TABLE OF CONTENTS | |
|---|---|---|
| 1. | SIGNATURE PAGE | 2 |
| 2. | TABLE OF CONTENTS | 3 |
| 3. | LIST OF ACRONYMS/ABBREVIATIONS | 4 |
| 4. | INTRODUCTION | 5 |
| 5. | STUDY OBJECTIVES | 5 |
| 5.1. | Primary Objective | 5 |
| 5.2. | Secondary Objectives | 5 |
| 6. | STUDY OVERVIEW | 5 |
| 7. | DEFINITIONS | 6 |
| 8. | ANALYSIS SET | 6 |
| 9. | STATISTICAL METHODS | 6 |
| 9.1. | General Principles | 6 |
| 9.1.1. | Handling Missing Values | 6 |
| 9.1.1.1. | Study Drug Administration Date or Time | 6 |
| 9.1.1.2. | Adverse Event or Concomitant Medications Dates or Times | 7 |
| 9.2. | Subject Disposition | 7 |
| 9.3. | Demographics and Baseline Characteristics | 7 |
| 9.3.1. | Demographics | 7 |
| 9.3.2. | Baseline Characteristics | 7 |
| 9.4. | Prior and Concomitant Medications | 8 |
| 9.5. | Study Drug Exposure | 8 |
| 9.6. | Efficacy Analysis | 8 |
| 9.7. | Health Economic Outcomes | 8 |
| 9.8. | Safety Analyses | 9 |
| 9.8.1. | Adverse Events | 9 |
| 9.8.2. | Vital Signs | 9 |
| 9.8.3. | Electrocardiograms | 9 |
| 9.8.4. | Physical examination | 9 |
| 9.8.5. | Clinical Laboratory | 9 |
| 9.8.6. | Other Analysis (urine drug screen, pregnancy test, alcohol breath test) | 9 |
| 9.9. | Pharmacokinetic Analysis | 9 |
| 10. | SAMPLE SIZE CALCULATIONS | 10 |
| 11. | TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES | 11 |
| 12. | TABLE OF CONTENTS FOR LISTING MOCK-UPS | 13 |

# 3. LIST OF ACRONYMS/ABBREVIATIONS

| Abbreviation | Description |
|--------------|---------------------------------------------------|
| AE | Adverse event |
| ATC | Anatomical therapeutic class |
| AUC | Area under the curve |
| BMI | Body mass index |
| CRF | Case report form |
| CSR | Clinical study report |
| d | days |
| ECG | Electrocardiogram |
| EMA | European Medicines Agency |
| ER | Emergency room |
| FDA | Food and Drug Administration |
| FSH | Follical stimulating hormone |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| IV | Intravenous |
| LIA | Local infiltration analgesia |
| LOS | Length of stay |
| MedDRA | Medical dictionary for regulatory affairs |
| min, m | minutes |
| MPADSS | Modified Post-Anesthesia Discharge Scoring System |
| n | Number of subjects |
| OBAS | Overall Benefit of Analgesia Score |
| OR | Operating room |
| PACU | Post-anesthesia care unit |
| PK | Pharmacokinetic(s) |
| PT | Preferred Term |
| NRS | Numeric rating scale |
| NRS-R | Numeric rating scale at rest |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SE | Standard error |
| SOC | System Organ Class |
| TEAE | Treatment-emergent adverse event |
| VAS | Visual analog scale |
| WHO-DD | World Health Organization – Drug Dictionary |
| WOCB | Women of child-bearing potential |
| yrs | years |

#### INTRODUCTION

This is a Phase 4, Multicenter, Randomized, Double-Blind, Controlled Study of EXPAREL for Postsurgical Pain Management in Subjects Undergoing Open Lumbar Spinal Fusion Surgery. Approximately 194 adult subjects undergoing primary, 1-2 level, open lumbar spinal fusion surgery under general anesthesia are planned for enrollment, in order to have at least 184 evaluable subjects.

This study was prematurely terminated by the sponsor. At the time of termination, the study has enrolled and treated 38 subjects.

The purpose of this SAP is to outline how the collected data will be summarized and presented for the abbreviated study report.

This SAP is developed based on

- Protocol 402-C-409 Amendment 2 issued on 2 August 2017.
- CRF version 1.0 issued on 30 September 2016.

The reader of this SAP is encouraged to also read the clinical protocol and other identified documents for details on the planned conduct of this study. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analyses.

#### 4. STUDY OBJECTIVES

#### 4.1. Primary Objective

The primary objective of this study is to compare postsurgical pain control following local infiltration analgesia (LIA) with EXPAREL admixed with bupivacaine HCl versus LIA with bupivacaine HCl in adult subjects undergoing open lumbar posterior spinal fusion surgery.

#### 4.2. Secondary Objectives

The secondary objectives of this study are to compare additional efficacy, safety, and health economic outcomes following LIA with EXPAREL admixed with bupivacaine HCl versus LIA with bupivacaine HCl in adult subjects undergoing open lumbar posterior spinal fusion surgery.

## 5. STUDY OVERVIEW

Subjects were screened within 30 days prior to study drug administration and at least one day prior to surgery. During the screening visit, subjects were assessed for past or present neurologic, cardiac, and general medical conditions that in the opinion of the Investigator would preclude them from study participation. After the informed consent form (ICF) was signed, a medical history, surgical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, clinical laboratory evaluations, urine drug screen, alcohol breath test, and urine pregnancy test for women of childbearing potential were collected (see Time and Events Schedule of Study Procedures in Section 12).

Subjects were randomized 1:1 to two treatment groups and stratified by surgery level (1-Level or 2-Level). Subjects in Group 1 received LIA with EXPAREL admixed with bupiviaine HCl and subjects in Group 2 received LIA with bupivacaine HCl.

## 6. **DEFINITIONS**

## Study Day

Study Day is calculated as the date of event minus the date of study drug administration plus one (1), if the date of event is on or after the date of study drug administration. Study Day equals the date of event minus the date of study drug administration if the date of event is before the date of study drug administration. Study days before the date of study drug administration will have negative values while those on or after the date of study drug administration are positive.

## Treatment-emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are AEs that occur after the administration of the study treatment through 30 days.

## Time 0 (zero)

Time 0 is defined as the date and time of the start of study drug administration.

#### Study Baseline

Study Baseline is defined as the last available measurement or assessment prior to the start of study drug administration.

#### 7. ANALYSIS SET

All Subjects: all the listings presented in this SAP will be based on all randomized subjects, unless specified otherwise.

## 8. STATISTICAL METHODS

## 8.1. General Principles

Only listings of subject data collected during the study will be provided. All listings will be sorted by treatment group, site ID, subject ID, and, if applicable, collection date and time.

## 8.1.1. Handling Missing Values

Data will be included in the listing as is. No imputed values will be included in the listings. However, in order to provide the drug safety profile, the missing or partial date/time will be imputed only for the determination of treatment emergency or prior/concomitant status.

#### 8.1.1.1. Study Drug Administration Date or Time

It is expected that all necessary information on study drug administration (start and stop date and time) will be complete. Any such information that is missing and cannot be obtained through

query resolution may be imputed, on a case-by-case basis, in a conservative manner that minimizes bias.

#### 8.1.1.2. Adverse Event or Concomitant Medications Dates or Times

For AEs or concomitant medications with missing or partially missing start/stop date/time, the following imputation rules will be applied when determining AE treatment-emergent status or medication prior/concomitant status:

For partial start date/time:

- If the year is unknown, then the date will be assigned as the date and time of first dose of study treatment.
- If the month is unknown, then:
  - i) If the year matches the year of study drug administration, then the month and day will be imputed to be the date and time of the first dose of study treatment.
  - ii) Otherwise, 'January' will be assigned.
- If the day is unknown, then:
  - i) If the month and year match the month and year of the dose of the study drug administration date, then the day will be imputed to be the day of study drug administration date.
  - ii) Otherwise, '01' will be assigned.
- If the time is unknown, then:
  - i) If the date (day, month, and year) matches the date of administration of study drug, then the time will be imputed to be the time of dose of study drug date.
  - ii) Otherwise, '00:00' will be assigned.

#### 8.2. Subject Disposition

A listing of subject disposition will be provided, which will include information on study completion status among others.

#### **8.3.** Demographics and Baseline Characteristics

#### 8.3.1. Demographics

Listing of demographic data will include:

- Age (years)
- Sex
- Ethnicity
- Primary Race

Age is presented as collected.

#### 8.3.2. Baseline Characteristics

Listing of baseline characteristic data will include:

• Height (cm)

#### Weight (kg) Body Mass Index (BMI) (kg/m²)

The formula for BMI is  $w/(h^2)$ , where w is weight in kilograms and h is height in meters. Weight in pounds will be converted to kilograms using the conversion factor of 2.2046 pounds to 1 kilogram. Height in inches will be converted to centimeters using the conversion factor of 2.54 centimeters to 1 inch. Height in centimeters will be converted to meters using the conversion factor of 100 centimeters to 1 meter.

#### 8.4. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD Sept. 2016 Enhanced) and will be classified according to the anatomical therapeutic chemical (ATC) classification system term (Level 4) and preferred name.

Prior medications are defined as medications with a stop date and time prior to the start of study drug administration.

Concomitant medications are defined as medications taken after the start of study drug administration (i.e., started prior to the start of study drug administration and continued after or started after the start of study drug administration).

Listing of prior and concomitant medications will include subject identification, treatment group, ATC class term and preferred name among others.

## 8.5. Study Drug Exposure

A listing of study drug exposure, which includes volume of injection administered, will be provided.

#### 8.6. Efficacy Analysis

Listing of the following efficacy assessments will be provided:

- -Pain intensity scores using the VAS
- -Pain Interference Scale (short form 6b)
- -Opioid rescue analgesics consumption
- -Treatment-emergent opioid-related AEs
- -OBAS questionnaire at 24, 48, and 72 hours or upon hospital discharge
- -Nurse's satisfaction with overall analgesia
- -Modified Postanesthesia Discharge Scoring System (MPADSS) criteria for discharge readiness

#### **8.7.** Health Economic Outcomes

Listing of the following health economic outcomes assessments done during the study will be provided: hospital length of stay (LOS), hospital readmissions, use of skilled nursing facility, and use of other health services following hospital discharge.

## 8.8. Safety Analyses

#### 8.8.1. Adverse Events

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 19.1 or later).

A treatment emergent adverse event (TEAE) is any adverse event with the onset date and time on or after the start date and time of study drug administration through postsurgical Day 30. Cardiac AEs of special interest include chest pain (angina, myocardial infarction), abnormal/irregular heart rate (bradycardia, tachycardia, extrasystoles), and shortness of breath requiring intervention. Neurologic AEs of special interest include altered mental status/altered sensorium, rigidity, dysarthria, seizure, tremors, metallic taste, tinnitus, perioral numbness, visual disturbance, and severe or worsening dizziness. In addition, the following events are of special interest if they persist or occur beyond 72-hours postdose: dizziness, hyperesthesia, muscular twitching, and tingling/paresthesia.

If an AE has a partial onset date and time the imputed start and stop dates and times will be used to determine treatment-emergence (e.g., an AE with stop date and time before the start date and time of study treatment is not treatment-emergent).

A listing of all AEs will be provided, with a flag indicating TEAEs.

#### 8.8.2. Vital Signs

Vital signs are resting heart rate (bpm), respiratory rate (beats per minute), oral body temperature (°C), systolic blood pressure (mmHg), and diastolic blood pressure (mmHg).

Listing of all vital signs collected at screening/Day 1 (pre-op) will be provided.

#### 8.8.3. Electrocardiograms

Data listings for ECG parameters collected at screening will be provided. The investigator's overall interpretation will be included.

#### 8.8.4. Physical examination

Listing of physical examination data collected at screening will be provided.

# 8.8.5. Clinical Laboratory

Listing of all clinical laboratory (hematology, chemistry, and urinalysis) tests collected at screening will be provided.

#### 8.8.6. Other Analysis (urine drug screen, pregnancy test, alcohol breath test)

A data listing of these will be provided.

#### 8.9. Pharmacokinetic Analysis

Drug concentrations are collected to assist the interpretation of adverse events. A data listing will be provided.

# 9. SAMPLE SIZE CALCULATIONS

The sample size was calculated based on VAS pain and total opioid results reported in Hughes et al (2016) and length of stay reported in the paper by Zheng et al (2002). Based on the reported efficacy for VAS pain intensity scores and assuming a 2-sided 0.05 alpha and a common SD of 70, a sample size of 50 subjects per treatment group should have at least 80% power to detect a 40-unit treatment difference. For total opioid consumption assuming a 2-sided 0.05 alpha and common standard deviation of the log-dose of 0.6 and 80% power a sample size of 64 subjects per treatment group is needed to detect a 30% difference in total opioid consumption through 48 hours. For length of stay assuming a 2-sided 0.05 alpha and common standard deviation of 2.4 and 80% power a sample size of 92 subjects per treatment group is needed to detect a 1 day difference in length of stay. Allowing for a 5% drop-outs rate a sample size of 97 subjects per treatment group should be enrolled to ensure 92 subjects provide length of stay data. A total study sample size of 184 evaluable subjects will provide 80% power to detect a 1-day difference in length of stay; 92% power to detect a 30% difference in total opioid consumption; and 97% power to detect a 40 point difference in VAS-AUC<sub>(0-72)</sub>.

# 10. TIME AND EVENTS SCHEDULE OF STUDY PROCEDURES

Pacira Pharmaceuticals, Inc.

402-C-409 (Spinal Fusion)

EXPAREL®

Clinical Study Protocol Amendment 2

Table 1. Time and Events Schedule of Study Procedures

| Visit Time Within With | Table 1. Time and Events Sched | die di St | Screen | D1 | 0 | | PACU | | | | | | | | Ī | | | | | | | D14 | D30 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Within Window 30 days | | | | | | OR | | 4h | бh | 8h | 10h | 12h | 24h | 28h | 32h | 36h | 48h | 52h | 56h | 60h | 72h | | |
| Window 30 days | | Time | Within | _ | | | | ±15 | ±30 | ±30 | | | | | | | | | | | | | |
| Assess/confirm eligibility Record medical and surgical history Record medical and surgical history X X² Conduct pregnancy test for WOCBP X X² Conduct pregnancy test for WOCBP X X² Conduct pregnancy test for WOCBP X X² Conduct truine drug screen X X X X X X X X X X X X X X X X X X X | | Window | 30 days | | | | | min | min | min | ±1h | ±1h | ±Ih | ±2h | ±2h | ±2h | ±2h | ±2h | ±2h | ±2h | ±4h | ±3d | ±3d |
| Record medical and surgical history X X X³ | Obtain signed ICF | | X | | | | | | | | | | | | | | | | | | | | |
| Record demographics and baseline characteristics | Assess/confirm eligibility | | X | Xa | | | | | | | | | | | | | | | | | | | |
| Conduct pregnancy test for WOCBP | Record medical and surgical history | | X | Xa | | | | | | | | | | | | | | | | | | | |
| Conduct urine drug screen | Record demographics and baseline characteristics | | X | | | | | | | | | | | | | | | | | | | | |
| Alcohol breath test X X X X X X X X X X X X X X X X X X X | Conduct pregnancy test for WOCBP | | X | | | | | | | | | | | | | | | | | | | | |
| Perform physical examination | Conduct urine drug screen | | X | Xª | | | | | | | | | | | | | | | | | | | |
| Measure vital signs (temperature, heart rate, respiratory rate and lood pressure) Measure vital signs (temperature, heart rate, respiratory rate and lood pressure) | Alcohol breath test | | X | | | | | | | | | | | | | | | | | | | | |
| A A A Science al labs (direct bilirubin and either GGT and LDH or ALT and AST) Perform 12-lead ECG Record VAS pain intensity score 1:23.4 Readomize subject, prepare study drug Administer scheduled presugical medications 3 Administer scheduled presugical medications 4 Administer study drug according to randomization schedule; record dart and stop times Record intraoperative opioids administered and doses Record surgery start and stop times Record surgery start and stop times Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics 1.5 Complete OBAS questionnaire 4 Nurse's satisfaction with postsurgical pain control 4 Pain Interference Scale Record date and time of actual discharge Document any hospital readmissions Document any hospital readmissions Document any unscheduled phone calls or office visits related to anin after discharge Record prior and concomitant medications 7 Record prior and concomitant medications 7 Record prior and concomitant medications 7 Record prior and concomitant medications 7 | Perform physical examination | | X | | | | | | | | | | | | | | | | | | | X | |
| Clinical labs (direct bilirubin and either GGT and LDH or ALT and AST) Record VAS pain intensity score <sup>1,23,4</sup> Randomize subject, prepare study drug Administer scheduled presurgical medications <sup>2</sup> Administer scheduled presurgical medications <sup>3</sup> Administer study drug according to randomization schedule; record tart and stop times Record intraoperative opioids administered and doses Record surgery start and stop times Record times and doses of all opioid rescue medication administered tart and stop times Complete OBAS questionnaire <sup>4</sup> Nurse's satisfaction with postsurgical pain control <sup>4</sup> Nain Interference Scale Record dime and time of actual discharge Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to to an after discharge Document any unscheduled phone calls or office visits related to an after discharge Document any unscheduled visits to the ER after discharge Document any unscheduled visits to the ER after discharge Na N | | ate and | X | Xª | | | | | | | | | | | | | | | | | | | |
| Record VAS pain intensity score <sup>1,2,3,4</sup> Randomize subject, prepare study drug Administer scheduled presurgical medications <sup>3</sup> X Administer scheduled presurgical medications <sup>3</sup> X Administer study drug according to randomization schedule; record tart and stop times Record surgery start and stop times Record surgery start and stop times Record surgery start and stop times Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics <sup>1,6</sup> Complete OBAS questionnaire <sup>4</sup> Nurse's satisfaction with postsurgical pain control <sup>4</sup> Ran Interference Scale Record date and time of actual discharge Document any hospital readmissions Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to sain after discharge Document any unscheduled visits to the ER after discharge | | r ALT and | X | | | | | | | | | | | | | | | | | | | | |
| Randomize subject, prepare study drug Administer scheduled presurgical medications <sup>3</sup> X Administer scheduled presurgical medications <sup>3</sup> X Administer study drug according to randomization schedule; record tart and stop times Record surgery start and stop times Record surgery start and stop times X Record times and doses of all opioid rescue medication administered administers cheduled postsurgical analgesics <sup>1,6</sup> Complete OBAS questionnaire <sup>4</sup> V Pain Interference Scale Record date and time of actual discharge Cocument any hospital readmissions Document use of skilled nursing facility Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to asin after discharge Record prior and concomitant medications <sup>7</sup> X X X X X X X X X X X X X | Perform 12-lead ECG | | X | | | | | | | | | | | | | | | | | | | | |
| Administer scheduled presurgical medications? Administer study drug according to randomization schedule; record tart and stop times Record intraoperative opioids administered and doses Record surgery start and stop times Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics. Complete OBAS questionnaire Nurse's satisfaction with postsurgical pain control Record date and time of actual discharge Document any hospital readmissions Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to sain after discharge Document any unscheduled visits to the ER after discharge Record prior and concomitant medications? | Record VAS pain intensity score <sup>1,2,3,4</sup> | | | X | | | X | X | Х | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Administer study drug according to randomization schedule; record that and stop times Record intraoperative opioids administered and doses Record surgery start and stop times Record times and doses of all opioid rescue medication administered Record times and topical analysesics. Record times of all opioid rescue medication administered X X X X X X X X X X X X X | Randomize subject, prepare study drug | | | X | | | | | | | | | | | | | | | | | | | |
| Record intraoperative opioids administered and doses Record surgery start and stop times Record surgery start and stop times Record surgery start and stop times Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics 1.6 Complete OBAS questionnaire 1 Nurse's satisfaction with postsurgical pain control 2 Pain Interference Scale Record date and time of actual discharge Cocument any hospital readmissions Cocument any hospital readmissions Cocument any unscheduled phone calls or office visits related to an after discharge Cocument any unscheduled visits to the ER after discharge Cocument any unscheduled visits to the ER after discharge Cocument and concomitant medications 7 Record prior and concomitant medications 7 | Administer scheduled presurgical medications <sup>5</sup> | | | X | | | | | | | | | | | | | | | | | | | |
| Record surgery start and stop times Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics 1.6 Complete OBAS questionnaire 4 Nurse's satisfaction with postsurgical pain control 4 Pain Interference Scale Record date and time of actual discharge Cocument any hospital readmissions Cocument use of skilled nursing facility Cocument any unscheduled phone calls or office visits related to pain after discharge Cocument any unscheduled visits to the ER after discharge Record prior and concomitant medications 7 Record prior and concomitant medications 7 | Administer study drug according to randomization sched<br>start and stop times | ule; record | | | Х | | | | | | | | | | | | | | | | | | |
| Record times and doses of all opioid rescue medication administered Administer scheduled postsurgical analgesics <sup>1,6</sup> Complete OBAS questionnaire <sup>4</sup> Nurse's satisfaction with postsurgical pain control <sup>4</sup> Pain Interference Scale X Record date and time of actual discharge Document any hospital readmissions Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to pain after discharge Record prior and concomitant medications <sup>7</sup> Record prior and concomitant medications <sup>7</sup> | Record intraoperative opioids administered and doses | | | | | Х | | | | | | | | | | | | | | | | | |
| Administer scheduled postsurgical analgesics 1.6 Complete OBAS questionnaire 4 Nurse is satisfaction with postsurgical pain control 4 Pain Interference Scale X Record date and time of actual discharge Cocument any hospital readmissions Cocument use of skilled nursing facility Cocument any unscheduled phone calls or office visits related to pain after discharge Cocument any unscheduled visits to the ER after discharge Record prior and concomitant medications 7 **The control of the | Record surgery start and stop times | | | | | Х | | | | | | | | | | | | | | | | | |
| Complete OBAS questionnaire <sup>4</sup> Nurse's satisfaction with postsurgical pain control <sup>4</sup> Pain Interference Scale X X X X X X X X X X X X X | Record times and doses of all opioid rescue medication a | dministered | | | | | ≪ | | | | | | | | | | | | | | | | > |
| Complete OBAS questionnaire <sup>4</sup> Nurse's satisfaction with postsurgical pain control <sup>4</sup> Pain Interference Scale X X X X X X X X X X X X X | Administer scheduled postsurgical analgesics 1,6 | | | | | | ⋖ | | | | | | | | | | | | | | - >- | | |
| Record date and time of actual discharge Cocument any hospital readmissions Cocument use of skilled nursing facility Cocument any unscheduled phone calls or office visits related to pain after discharge Cocument any unscheduled visits to the ER after discharge Record prior and concomitant medications X X X X X X X X X X X X X | Complete OBAS questionnaire <sup>4</sup> | | | | | | | | | | | | X | | | | Х | | | | X | | |
| Record date and time of actual discharge Document any hospital readmissions Cocument use of skilled nursing facility Cocument any unscheduled phone calls or office visits related to pain after discharge Cocument any unscheduled visits to the ER after discharge Record prior and concomitant medications X X X X X | Nurse's satisfaction with postsurgical pain control <sup>4</sup> | | | | | | | | | | | | X | | | | X | | | | Х | | |
| Document any hospital readmissions Document use of skilled nursing facility Document any unscheduled phone calls or office visits related to pain after discharge Document any unscheduled visits to the ER after discharge Record prior and concomitant medications X X X | Pain Interference Scale | | | X | | | | | | | | | | | | | | | | | | X | |
| Document any hospital readmissions Cocument use of skilled nursing facility Cocument any unscheduled phone calls or office visits related to pain after discharge Cocument any unscheduled visits to the ER after discharge Record prior and concomitant medications X X X X X | Record date and time of actual discharge | | | | | | | | | | | | | | | | ⋖. | | | | | > | |
| Document any unscheduled phone calls or office visits related to pain after discharge Document any unscheduled visits to the ER after discharge Record prior and concomitant medications X X X | Document any hospital readmissions | | | | | | | | | | | | | | | | | | | | | X | X |
| pain after discharge Document any unscheduled visits to the ER after discharge Record prior and concomitant medications **T A A A A A A A A A A A A A A A A A A | Document use of skilled nursing facility | | | | | | | | | | | | | | | | | | | | | X | X |
| Document any unscheduled visits to the ER after discharge XX X Record prior and concomitant medications X X X | | lated to | | | | | | | | | | | | | | | | | | | | v | v |
| Record prior and concomitant medications | pain after discharge | | | | | | | | | | | | | | | | | | | | | | |
| | | ge | | | | | | | | | | | | | | | | | | | | X | X |
| Record AEs (beginning at the time ICF is signed) <sup>8</sup> | Record prior and concomitant medications | | ≪ | | | | | | | | <del> </del> | | | | | | | | | | | | >- |
| | Record AEs (beginning at the time ICF is signed) <sup>8</sup> | | <b>▼</b> | | | | | | | | <u> </u> | | | | | | | | | | | | - > |

CONFIDENTIAL Page 11 of 44 5 March 2018

Abbreviations: AE = adverse event; ALT = alanine transaminase; AST = aspartate transaminase; d = day; D = day; ECG = electrocardiogram; ER = emergency room; GGT=Gamma-glutamyl transpeptidase; h = hours; ICF = informed consent form; LDH = lactate dehydrogenase; min = minutes; OBAS = overall benefit of analgesia score; OR = operating room; PACU = post-anesthesia care unit; Preop = preoperative; q12h = every 12 hours; VAS = visual analog scale; WOCBP = women of childbearing potential.

- a: If the Screening Visit is conducted within 10 days of the date of surgery, the following Day-1 pre-op assessments are not required: assess/confirm eligibility; record medical and surgical history; conduct pregnancy test for WOCBP; conduct urine drug screen; and measure vital signs (temperature, heart rate, respiratory rate and blood pressure)
- \* Postsurgical assessments will be conducted at the timepoints specified after the end of surgery. All assessments conducted after baseline (ie, study drug administration) will be timed from the end of surgery, defined as the time of last suture/staple. At timepoints when multiple assessments coincide, the VAS pain intensity assessment will be conducted first.
- Timepoints shown through 72 hours. Note: if discharge occurs before 72 hours, the study coordinator must stress to the patient the importance of completing the scheduled pain intensity assessments up to 72 hours. These assessments should be recorded by the patient in the patient log provided upon discharge.
- 2 The preoperative pain intensity assessment should be conducted prior to administration of any premedication.
- 3 Also record VAS pain intensity scores immediately prior to each administration of rescue pain medication, and just prior to hospital discharge.
- 4 And just prior to hospital discharge. Note: if discharge occurs before 72 hours, the study coordinator must stress to the patient the importance of completing the scheduled OBAS questionnaire up to 72 hours. Completion of the questionnaire should be recorded by the patient in the patient log provided upon discharge.
- 5 Administer presurgical analgesics (ie, acetaminophen 975-1000 mg orally (PO), celecoxib 200 mg PO [or naproxen 500 mg PO twice a day or meloxicam 7.5 mg PO once a day in case of allergy], and gabapentin up to 900 mg PO).
- 6 Administer scheduled post-surgical analgesics (ie, acetaminophen 975-1000 mg PO every 8 hours (q8h) [maximum of 3000 mg per day; acetaminophen IV can be used if the patient is unable to tolerate oral acetaminophen], celecoxib 200 mg PO every 12 hours up to 48 hours (q12h; or naproxen 500 mg PO twice a day or meloxicam 7.5 mg PO once a day in case of allergy), cyclobenzaprine 10 mgq8h, and gabapentin up to 900 mg PO q8h).
- 7 Instruct subject to discontinue prohibited medications. Record date and time of all medications starting at least 30 days prior to study drug administration until hospital discharge. Record medications administered for treatment of an AE through Day 30.
- If a cardiac AE (eg, chest pain [angina, myocardial infarction], abnormal/irregular heart rate [bradycardia, tachycardia, extrasystoles], or shortness of breath), neurological AE (eg, altered mental status/altered sensorium, dizziness, dysarthria, hyperesthesia, metallic taste, peroral numbness, seizure, tinnitus, tremors, visual disturbance, muscular twitching or rigidity beyond 72 hours postdose, or tingling/paresthesia beyond 72 hours postdose), or serious AE (SAE) occurs during the study, a 12-lead ECG, vital signs, PK draw, and any appropriate clinical laboratory tests should be conducted as close as possible to when the event occurs.

CONFIDENTIAL Page 12 of 44 5 March 2018

# 11. TABLE OF CONTENTS FOR LISTING MOCK-UPS

| LISTING | 16.1-7: RANDOMIZATION - ALL SUBJECTS | 15 |
|---|---|---|
| LISTING | 16.2-1: SUBJECT DISPOSITION | 16 |
| LISTING | 16.2-2: DEMOGRAPHICS - ALL SUBJECTS | 17 |
| LISTING | 16.2-3: BASELINE CHARACTERISTICS - ALL SUBJECTS | 18 |
| LISTING | 16.2-4: PROTOCOL DEVIATION - ALL SUBJECTS | 19 |
| LISTING | 16.2-5: INCLUSION/EXCLUSION CRITERIA - ALL SUBJECTS | 20 |
| LISTING | 16.2-6: MEDICAL HISTORY - ALL SUBJECTS | 21 |
| LISTING | 16.2-7: STUDY DRUG EXPOSURE - ALL SUBJECTS | 22 |
| LISTING | 16.2-8: VISITS - ALL SUBJECTS | 23 |
| LISTING | 16.2-9.1: ADMISSION AND DISCHARGE - ALL SUBJECTS | 24 |
| LISTING | 16.2-9.2: SURGERY - ALL SUBJECTS | 25 |
| LISTING | 16.2-10: PAIN INTENSITY - VISUAL ANALOG SCALE - ALL SUBJECTS | 26 |
| LISTING | 16.2-11: PAIN INTERFERENCE | 27 |
| LISTING | 16.2-12: DISCHARGE READINESS - ALL SUBJECTS | 28 |
| LISTING | 16.2-13: NURSE SATISFACTION - ALL SUBJECTS | 29 |
| LISTING | 16.2-14: OBAS QUESTIONNAIRE - ALL SUBJECTS | 30 |
| LISTING | 16.2-15: LAST PHONE CALL - ALL SUBJECTS | 31 |
| LISTING | 16.2-16.1: ALL ADVERSE EVENTS | 32 |
| LISTING | 16.2-16.2: ALL SERIOUS ADVERSE EVENTS - ALL SUBJECTS | 32 |
| LISTING | 16.2-16.3: TREATMENT-EMERGENT SERIOUS ADVERSE EVENTS - ALL SUBJECTS | 33 |
| LISTING | 16.2-16.4: TREATMENT-EMERGENT SERIOUS ADVERSE EVENTS LEADING TO STUDY DISCONTINUATION - ALL SUBJECTION - ALL | TS<br>33 |
| LISTING | 16.2-16.5: TREATMENT-EMERGENT OPIOID-RELATED ADVERSE EVENTS - ALL SUBJECTS | 33 |
| LISTING | 16.2-16.6.1: CARDIAC TREATMENT-EMERGENT ADVERSE EVENTS OF SPECIAL INTEREST - ALL SUBJECTS | 33 |
| LISTING | 16.2-16.6.2: NEUROLOGIC TREATMENT-EMERGENT ADVERSE EVENTS OF SPECIAL INTEREST - ALL SUBJECTS | 33 |
| LISTING | 16.2-17: PHARMACOKINETICS - ALL SUBJECTS | 34 |
| LISTING | 16.2-18: VITAL SIGNS ASSESSMENT - ALL SUBJECTS | 35 |
| LISTING | 16.2-19.1: CONCOMITANT MEDICATIONS - ALL SUBJECTS | 36 |

| Pacira Pharmaceuticals, Inc. EXPAREL | 402-C-409<br>Statistical Analysis Plan |
|---|---|
| LISTING 16.2-19.2: PRIOR MEDICATIONS - ALL SUBJECTS | 36 |
| LISTING 16.2-19.3: INTRAOPERATIVE OPIOIDS - ALL SUBJECTS | 37 |
| LISTING 16.2-19.4: RESCUE MEDICATION - ALL SUBJECTS | 37 |
| LISTING 16.2-20: ELECTROCARDIOGRAM FINDINGS - INVESTIGATOR ASSESSMENT - ALL SUBJECTS | 38 |
| LISTING 16.2-21: PHYSICAL EXAMINATION | 39 |
| LISTING 16.2-22: URINE DRUG SCREEN - ALL SUBJECTS | 40 |
| LISTING 16.2-23: PREGNANCY TEST FOR WOMEN OF CHILD BEARING POTENTIAL | 41 |
| LISTING 16.2-24: CLINICAL LABORATORY TESTS-HEMATOLOGY - ALL SUBJECTS | 42 |
| LISTING 16.2-25: CLINICAL LABORATORY TESTS-CHEMISTRY - ALL SUBJECTS | 42 |
| LISTING 16.2-26: CLINICAL LABORATORY TESTS-URINALYSIS - ALL SUBJECTS | 42 |
| LISTING 16.2-27: UNIQUE ADVERSE EVENTS TERMS AND ASSOCIATED CODED TERMS | 43 |
| LISTING 16.2-28: UNIQUE MEDICATION TERMS AND ASSOCIATED CODED TERMS | 44 |

Protocol: 402-C-409

Pacira Pharmaceuticals
Listing 16.1-7: Randomization - All Subjects

(Page X of Y)

| | | | Randomi | zation | | | |
|---|---|---|---|---|---|---|---|
| Subject | Site<br>Number | Date/ Day[1] | Time | Number | Treatment | Surgery<br>type | Screw<br>type |
| XXX-YYYY | XXX | yyyy-mm-dd/ xxx | hh:mm | XXXXX | XXXXXX | 2-Level | pedicle |

[1]Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 1-7.sas

DateTime

Note to programmer: Analysis set will by 'Y' if subject in set, blank otherwise.

| Pacira Pharmaceuticals, Inc. | 402-C-409 |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-1: Subject Disposition - All Subjects

| Treatment: | | | | | | |
|---|---|---|---|---|---|---|
| | Informed | | First | Last | End of | |
| | Consent | Randomization | Dose | Visit | Study | Primary Reason for |
| Subject | Date/ Day[1] | Date/ Day[1] | Date/ Day[1] | Date/ Day[1] | Status | Early Termination |
| XXX-YYYY | yyyy-mm-dd/ xxx | yyyy-mm-dd/ xxx | yyyy-mm-dd/ xxx | yyyy-mm-dd/ xxx | Completed | Study Terminated By Sponsor |

[1]Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-1.sas

DateTime

Note to programmer: End of study status for subject who early terminated from the study is the primary reason for termination. If subject discontinued due to an AE then the reason should read 'ADVERSE EVENT, AE # X'. If subject discontinued due to death the reason should read 'DEATH ON DDMONYYYY'. For those reasons that also collected a specify text, concatenate into "Primary Reason" as "Other, Specify: ...".

| Pacira Pharmaceuticals, Inc. | 402-C-409 |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

| Pacira Pharmaceuticals Listing 16.2-2: Demographics - All Subjects | | | | S | (Page X of Y | 7) | | Prot | ocol: 402-C-409 |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | : | | | | | | | | |
| | Subject | | Age | | Child Bearing | | | ASA | |
| Subject | Initials | Birth Date | (yrs) | Sex | Potential? | Primary Race | Ethnicity | Class | Country |
| | | | | | | | | | <u>.</u> |

XXXXXXXXXXXXXXXX XXXXXXX

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-2.sas

XXX-YYYY AMZ yyyy-mm-dd XX XXXXXX

DateTime

XXXXXXX

Note to programmer: If Primary Race is 'other' then Primary Race should be 'Other: other-specify-text'.

| Pacira Pharmaceuticals, Inc. | 402-C-409 |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409

Listing 16.2-3: Baseline Characteristics - All Subjects

Treatment:

| rreatment: | | | | Body Mass Index |
|------------|------------------|-------------|-------------|-----------------|
| Subject | Date | Height (cm) | Weight (kg) | (kg/m²) |
| XXX-YYYY | yyyy-mm-ddThh:mm | XXX.X | XXX.X | XX.X |

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-3.sas

| Pacira Pharmaceuticals, Inc. | 402-C-409 | |
|---|---|---|
| EXPAREL | Statistical Analysis Plan | |
| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |

| Treatment: | | | | | | |
|---|---|---|---|---|---|---|
| Subject | Date of<br>Deviation /<br>Day[1] | Time of<br>Deviation | Deviation Type | Deviation<br>Description | Action Taken | If Other, specify |
| XXX-YYYY | yyyy-mm-dd/ xxx | Thh:mm | Study Drug Error | xxxxxxxxxxxxx | Staff Retraining | |

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-4.sas

Listing 16.2-4: Protocol Deviation - All Subjects

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

| Pacira Pharr<br>EXPAREL | maceuticals, Inc. | | 402-C-409<br>Statistical Analysis Plan | |
|---|---|---|---|---|
| | narmaceuticals 6.2-5: Inclusion | Exclusion Crite | X of Y) | Protocol: 402-C-409 |
| Treatment | Met all | | | |
| Subject | eligibility criteria? | Category | Criterion ID<br>Failed | Protocol Version<br>Enrolled under |
| | | <u> </u> | | |
| XXX-YYYY | No | Exclusion | | Original |

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-5.sas

| Pacira Ph | armaceuticals (Page X of | Y) | | Protocol: 402-C-409 |
|---|---|---|---|---|
| Listing 1 | 6.2-6: Medical History - All Subjects | | | |
| Treatment | : | | | |
| | V: Verbatim Term | | | |
| Subject | S: System Organ Class[1] | Start | Stop | |
| ID | P: Preferred Term[1] | Date | Date | |
| xxx-xxxx | V: vvvvvvvvvvvvvvvvvvv | YYYY-MM-DD | YYYY-MM-DD | |
| | S: ssssssssssssssssss | | | |
| XXX-XXXX | P: pppppppppppppppppp | | | |
| xxx-xxxx | V: vvvvvvvvvvvvvvvvvvvv | YYYY | Ongoing | |
| | S: ssssssssssssssssss | | | |
| xxx-xxxx | P: ppppppppppppppppp | | | |
| xxx-xxx | V: vvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvv | YYYY-MM-DD | Ongoing | |
| | S: ssssssssssssssssssssssss | | | |
| xxx-xxxx | P: pppppppppppppppppppppppppppppppppppp | | | |
| | V: vvvvvvvvvvvvvvvvvvvv | YYYY-MM | Ongoing | |
| | S: sssssssssssssssssssssssssssss | | | |
| | P: ppppppppppppppppp | | | |
| xxx-xxxx | V: vvvvvvvvvvvvvvvvvvvvvvvvvvv | YYYY-MM-DD | YYYY-MM-DD | |
| | S: sssssssss | | | |
| | P: ppppppppppp | | | |

Programming note: For subjects with multiple records, present in the order of onset date.

Source: list SAS datasets used to create table M:\402C409\production\programs\t1f\ $L16_2-6.sas$  DateTime

<sup>[1]</sup> MedDRA vxx.x.

| Pacira Pharmaceuticals, Inc. |
|------------------------------|
| EXPAREL |

402-C-409 Statistical Analysis Plan

Protocol: 402-C-409

Pacira Pharmaceuticals Listing 16.2-7: Study Drug Exposure - All Subjects (Page X of Y)

| Treatment: | | | | |
|------------|-----------------|-------|-------|--------------|
| | | Start | Stop | Total Volume |
| Subject | Date/ Day[1] | Time | Time | (mL) |
| XXX-YYYY | vvvv-mm-dd/ xxx | HH:MM | HH:MM | XXX |

[1] Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-7.sas$ 

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409
Listing 16.2-8: Visits - All Subjects

| Treatment | : | |
|-----------|------------|--------------------|
| Subject | Visit | Visit Date/ Day[1] |
| XXX-YYYY | Screening | yyyy-mm-dd/ xxx |
| | D1 (Preop) | yyyy-mm-dd/ xxx |
| | D14 | yyyy-mm-dd/ xxx |
| | D30 Call | yyyy-mm-dd/ xxx |

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-8.sas$ 

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409

Listing 16.2-9.1: Admission and Discharge - All Subjects
Treatment:

| Subject | Date of admission to surgical facility/ Day[1] | Time of admission to surgical facility | Date of admission to PACU/ Day[1] | Time of admission to PACU | Date of discharge from surgical facility/ Day[1] | Time of discharge from surgical facility |
|---|---|---|---|---|---|---|
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | yyyy-mm-dd/ xxx | hh:mm | yyyy-mm-dd/ xxx | hh:mm |

[1] Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-9\_1.sas

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |
|---|---|---|
| Listing 16.2-9.2: Surgery - All Subjects | | |

Treatment:

| Subject | Date/ Day[1] | Start<br>Time | End<br>Time | Procedure<br>Name | Level of<br>Surgery | Surgery<br>performed by | Total<br>Incision<br>Length | Type of Anesthesia | Intraoperative opioids administered? |
|---|---|---|---|---|---|---|---|---|---|
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | hh:mm | | | | | Other:xxx_specify_ | No |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | hh:mm | | | | | | |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | hh:mm | | | | | | |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | hh:mm | | | | | | |

[1] Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-9 2.sas

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-10: Pain Intensity - Visual Analog Scale - All Subjects

Treatment:

| Subject | Date/ Day[1] | Timepoint | Time | Pain assessment [2] |
|----------|-----------------|--------------|-------|---------------------|
| XXX-YYYY | yyyy-mm-dd/ xxx | PACU Arrival | hh:mm | XXX |
| | yyyy-mm-dd/ xxx | 4 Hours | hh:mm | XXX |
| | yyyy-mm-dd/ xxx | 6 Hours | hh:mm | XXX |
| | yyyy-mm-dd/ xxx | 8 Hours | hh:mm | XXX |

. . .

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-10.sas

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

<sup>[2]</sup> How much pain are you experiencing right now (in VAS, cm)?

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-11: Pain Interference - All Subjects

Treatment:

| Subject | Date/ Day[1] | Timepoint | Question | Res<br>ponse[2] |
|---|---|---|---|---|
| | | | In the past seven days, | |
| XXX-YYYY | yyyy-mm-dd/ xxx | 24 Hours | 1. How much did pain interfere with your enjoyment of life? | 2 |
| | | | 2. How much did pain interfere with your ability to concentrate? | 1 |
| | | | 3. How much did pain interfere with your day to day activities? | 1 |
| | | | 4. How much did pain interfere with your enjoyment of recreational | |
| | | | activities | 4 |
| | | | 5. How much did pain interfere with doing your tasks away from home? | 5 |
| | | | 6. How often did pain keep you from socializing with others? | 3 |

. . .

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-11.sas

*DateTime* 

Note to programmer: Sort by date and time within subject.

Continue for Timepoint = 48 Hours, 72 Hours

<sup>[1]</sup>Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

<sup>[2]</sup> For questions 1 to 5, 1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, 5 = Very much. For question 6, 1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always.

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |
|---|---|---|
| Listing 16.2-12: Discharge Readiness - All Subjects | | |
| Treatment · | | |

| Subject | Timepoint | Date/ Day[1] | Time | Vital<br>Sign[2] | Ambu<br>Lation[3] | Nausea and Vomiting[4] | | Surgical<br>Bleeding[4<br>] |
|---|---|---|---|---|---|---|---|---|
| XXX-YYYY | Day of Surgery | yyyy-mm-dd/ xxx | hh:mm | 2 | 1 | 0 | 1 | 2 |

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-12.sas$ 

DateTime

#### Note to programmer:

Sort by date and time within subject.

Continue for Timepoint = Day 2 Morning, Day 2 Evening, Discharge

<sup>[2]</sup> 2 = <=20% of preoperative value, 1 = 20%-40% of preoperative value, 0 = >40% of preoperative value

<sup>[3] 2 =</sup> Steady gait/no dizziness, 1 = With assistance, 0 = None/dizziness

<sup>[4] 2 =</sup> Minimal, 1 = Moderate, 0 = Severe

Pacira Pharmaceuticals, Inc.

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409

Listing 16.2-13: Nurse Satisfaction - All Subjects Treatment:

| Subject | Date/ Day[1] | Time | Timepoint | Nurse's Overall<br>Satisfaction [2] |
|---|---|---|---|---|
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | 24 Hours | 2 |

. . .

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-13.sas

DateTime

#### Note to programmer:

Sort by date and time within subject.

Continue for Timepoint = 48 Hours, 72 Hours

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

<sup>[2]</sup> Nurse's overall satisfaction with the pain medication received after surgery:

<sup>1 =</sup> Extremely dissatisfied, 2 = Dissatisfied, 3 = Neither satisfied nor dissatisfied,

<sup>4 =</sup> Satisfied, 5 = Extremely satisfied

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409

Listing 16.2-14: OBAS Questionnaire - All Subjects
Treatment:

| | | | | | Res |
|---|---|---|---|---|---|
| Subject | Date/ Day[1] | Time | Timepoint | Question | ponse |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | 24 Hours | <ol> <li>Was the OBAS Questionnaire Completed?</li> <li>Please rate your current pain at rest</li> <li>Please grade any distress and bother from vomiting in the past 24 h</li> <li>Please grade any distress and bother from itching in the past 24 h</li> <li>Please grade any distress and bother from sweating in the past 24 h</li> <li>Please grade any distress and bother from freezing in the past 24 h</li> <li>Please grade any distress and bother from dizziness in the past 24 h</li> <li>How satisfied are you with your pain treatment during the past 24 h</li> <li>Number of days in the Nursing Facility</li> </ol> | |

[1]Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\ 2-14.sas$ 

DateTime

Note to programmer: Sort by date and time within subject.

Continue for Timepoint = 48 Hours, 72 Hours

Pacira Pharmaceuticals Protocol: 402-C-409 (Page X of Y) Listing 16.2-15: Last Phone Call - All Subjects

Treatment:

| Subject | Date/ Day[1] | Question | Response |
|---|---|---|---|
| XXX-YYYY | yyyy-mm-dd/ xxx | 1. Was Day 29 Phone Call made to the subject? | Yes |
| | | 2. Were there any unscheduled pain-related calls since subject discharge? | Yes |
| | | 3. Number of pain-related phone calls | 2 |
| | | 4. Were there any unscheduled pain-related visits since subject discharge? | No |
| | | 5. Number of pain-related office visits | 0 |
| | | 6. Were there any Emergency Department Visits since subject discharge? | Yes |
| | | 7. Number of Emergency Department Visits | 1 |
| | | 8. Was there any Skilled Nursing Facility admission since subject discharge? | No |
| | | 9. Number of days in the Nursing Facility | 0 |
| | | 10. Was there any hospital readmission since subject discharge? | No |
| | | 11. Number of hospital readmission | 0 |

[1] Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table  $M: \402C409\production\programs\tlf\Ll6_2-15.sas$ 

DateTime

402-C-409

Note to programmer: Sort by date within subject.

| Pacira Pharmaceuticals Listing 16.2-16.1: All Adverse Events - All S | | | ll Su | ıbj∈ | (Page X of Y) | Protocol: 402-C-409 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatmernt: | | | | | | | | | | |
| Subject<br>ID | Start<br>Date/<br>Day[1] | Stop<br>Date/<br>Day[1] | Duration<br>(Day)[2] | TEAE | S: | Verbatim<br>System Organ Class[3]<br>Preferred Term[3] | S: Severity<br>R: Relationship<br>SAE: Serious | F: Frequency A: Action Taken O: Outcome | I: | AESI |
| xxxxx | YYYY-MM-DD/<br>XXX | YYYY-MM-DD/<br>XXX | ′ XXX | Yes | s: | vvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvv | S: Moderate<br>R: Not Related<br>SAE: Death | F: xxx<br>A: Hospitalization<br>O: Fatal | | |
| | YYYY-MM-DD/<br>XXX | YYYY-MM-DD/<br>XXX | ′ XXX | Yes | S: | vvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvv | S: Mild<br>R: Possible<br>SAE: Life<br>Threatening | F: xxx<br>A: Study Drug Disc<br>O: Recovered | | |
| xxxxx | YYYY-MM-DD/<br>XXX | YYYY-MM-DD/<br>XXX | ′ XXX | No | s: | vvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvv | S: Severe<br>R: Probable<br>SAE: Incapacity | F: xxx<br>A: Nonpharm Therapy<br>O: Recovered with<br>Sequelae | | |
| | YYYY-MM-DD/<br>XXX | | | Yes | S: | vvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvvv | S: Severe<br>R: Definite<br>SAE: Hospital | F: xxx<br>A: Other: xxx<br>O: Not Recovered | | |
| Program | nming instruct | tions: Sort | by Subjec | ct ID | | hen Start Date. | SAL. MOSPICAL | o. Not Recovered | | |

TEAE: Treatment-emergent AE (Yes=TEAE/No=Not TEAE)

[1] Day=event date - first dose date +1 if event occurred on/after first dose; Otherwise Day=event date - first dose date.

- [2] Duration=Stop Date Start Date +1.
- [5] MedDRA version 19.0.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-16\_1.sas

DateTime

**Note to programmer:** If AE is ongoing, put ONGOING in stop row. Do not split an AE across pages. Insert a page break between subjects.
Use this mock-up for the following listings:

Listing 16.2-16.2: All Serious Adverse Events - All Subjects

```
Listing 16.2-16.3: Treatment-emergent Serious Adverse Events - All Subjects
Listing 16.2-16.4: Treatment-emergent Serious Adverse Events leading to study discontinuation - All Subjects
Listing 16.2-16.5: Treatment-emergent Opioid-Related Adverse Events - All Subjects
Listing 16.2-16.6.1: Cardiac Treatment-emergent Adverse Events of Special Interest - All Subjects
Listing 16.2-16.6.2: Neurologic Treatment-emergent Adverse Events of Special Interest - All Subjects
```

#### Note:

Cardiac AEs of special interest include chest pain (angina, myocardial infarction), abnormal/irregular heart rate (bradycardia, tachycardia, extrasystoles), and shortness of breath requiring intervention. Neurologic AEs of special interest include altered mental status/altered sensorium, rigidity, dysarthria, seizure, tremors, metallic taste, tinnitus, perioral numbness, visual disturbance, and severe or worsening dizziness. In addition, the following events are of special interest if they persist or occur beyond 72-hours postdose: dizziness, hyperesthesia, muscular twitching, and tingling/paresthesia.

| Pacira Pharmaceuticals, Inc. | 402-C-409 |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |
|---|---|---|
| Listing 16 2-17. Pharmacokinetics - All Subjects | | |

Treatment:

| Subject | Collection Date/ Day[1] | Collection<br>Time | Vaule | Reason for PK<br>Collection | If Other, Specify |
|---|---|---|---|---|---|
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm hh:mm hh:mm hh:mm | xxx<br>xxx<br>xxx | AE Special Interest<br>Other<br>SAE | xxxxxxxxxxx |

. . .

. . .

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-17.sas$ 

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Protocol: 402-C-409

Pacira Pharmaceuticals (Page X of Y)

Listing 16.2-18: Vital Signs Assessment - All Subjects

Treatment:

| | | | | Heart | Oral | Blood Pres | sure (mmHg) |
|---|---|---|---|---|---|---|---|
| Subject | Date/ Day[1] | Time | Timepoint | Rate<br>(bpm) | Temperature<br>(°C) | Systolic | Diastolic |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm<br>hh:mm | Screening<br>Day 1 (Pre-op) | XX<br>XX | XX.X<br>XX.X | XXX<br>XXX | XX<br>XX |

[1] Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-18.sas

DateTime

Note to programmer: Sort by date and time within subject.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409

Listing 16.2-19.1: Concomitant Medications - All Subjects

| Treatment | t: | | | |
|---|---|---|---|---|
| | Start Date | V: Verbatim | D: Dose & Unit | Indication |
| | (day) [1] | D: Generic Name[2] | R: Route & Form | AE: AE number |
| Subject | Stop Date | C: Medication Class[2] | F: Frequency | MH: Medical History |
| ID | (day) [1] | | | _ |
| XXXXX | YYYY-MM-DD (XX) | V: mmmmmmmmmmmmmm | D: dddddddd uuuuuuu | AE: xx |
| | Continuing | D: nnnnnnnnnnnnnn | R: rrrrrrr | |
| | | C: ppppppppppp | F: ffffffff | |
| XXXXX | YYYY-MM-DD (XX) | V: mmmmmmmmmmmmmm | D: dddddddd uuuuuuu | MH: Hypertension |
| | YYYY-MM-DD (XX) | D: nnnnnnnnnnnnnn | R: rrrrrrr | |
| | | C: ppppppppppp | F: ffffffff | |
| | YYYY-MM-DD (XX) | V: mmmmmmmmmmmmm | D: dddddddd uuuuuuu | Prophylactic |
| | , , | | | riophylactic |
| | YYYY-MM-DD (XX) | D: nnnnnnnnnnnnnn | R: rrrrrrr | |
| | | C: ppppppppppp | F: ffffffff | |
| xxxxx | YYYY | V: mmmmmmmmmmmmmmmmmmmmmmmmmmmmmmmmmmmm | D: dddddddd uuuuuuu | aaaaa bbbbbb ccccc |
| | Continuing | D: nnnnnnnnnnnnnn | R: rrrrrrr | |
| | Concentating | C: ppppppppppp | F: fffffff | |
| | | •• | | |
| | YYYY-MM | V: mmmmmmmmmmmmm | D: dddddddd uuuuuuu | aaaaa bbbbbb ccccc |
| | Continuing | D: nnnnnnnnnnnnnn | R: rrrrrrr | |
| | , and the second | C: ppppppppppp | F: ffffffff | |

Programming note: Display 'Ongoing' for Stop Date if stop date is missing and the Ongoing tick box is checked. Within a subject, medications should be presented in order of earliest start date. Do not display day for incomplete dates. If Reason for Use is 'Prophylactic', display 'Prophylactic' in the respective Indication cell. If unit, route, and frequency is other, include other specify text

- [1] Day = Medication date First dose date + 1.
- [2] Preferred Term and ATC4, WHODD version xxx.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-19 1.sas

DateTime

Listing 16.2-19.2: Prior Medications - All Subjects

Replace foonote [1] with "Day = Medication date - First dose date"

Listing 16.2-19.3: Intraoperative Opioids - All Subjects

Listing 16.2-19.4: Rescue Medication - All Subjects

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-20: Electrocardiogram Findings - Investigator Assessment - All Subjects

| Treatment: | | | | |
|---|---|---|---|---|
| | Assessment | Assessment | | |
| Subject | Date/ Day[1] | Time | Visit | Finding Specify |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | Screening | Normal |
| XXX-YYYY | yyyy-mm-dd/ xxx | hh:mm | Screening | Abormal-CS xxxxxxxxxx |

[1]Day=Visit date - first dose date +1 if Visit is on/after first dose date; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-20.sas

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-21: Physical Examination - All Subjects

Treatment:

| Subject | Visit | Assessment Date /Day[1] | Assessment<br>time | Body System | Condition | Abnormality |
|---|---|---|---|---|---|---|
| XXX-YYYY | Screening | yyyy-mm-dd/ xxx | hh:mm | General Appearance | Normal | |
| | | | | HEENT | Abnormal | L thyroid mass-<br>2x3cm; immobile,<br>nontender; NCS |
| | | | | Cardiovascular | Normal | |
| | | | | Bronchopulmonary | No Change | |
| | | | | Abdomen/Gastrointestinal | Normal | |
| | | | | Lymphatic | Normal | |
| | | | | Musculoskeletal | Normal | |
| | | | | <pre>Integumentary (skin, hair, nails, etc.)</pre> | Normal | |
| | | | | Neurologic | Normal | |
| | | | | Extremities | Normal | |

[1]Day=Visit date - first dose date +1 if Visit is on/after first dose date; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-21.sas

| Pacira Pharmaceuticals, Inc. | 402-C-409 |
|------------------------------|---------------------------|
| EXPAREL | Statistical Analysis Plan |

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |
|---|---|---|
| Listing 16 2-22: Urine Drug Screen - All Subjects | | |

Treatment:

| Subject | Timepoint | Date/ Day[1] | Time | Specimen<br>Type | Result |
|----------|-----------|-----------------|-------|------------------|----------|
| XXX-YYYY | Screening | yyyy-mm-dd/ xxx | hh:mm | Urine | Negative |

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-22.sas$ 

DateTime

#### Note to programmer:

Sort by date and time within subject.

| Pacira Pharmaceuticals | (Page X of Y) | Protocol: 402-C-409 |
|---|---|---|
| Listing 16.2-23: pregnancy test for | Women of Child Bearing Potential - All Subjects | |
| Treatment: | | |

| Subject | Timepoint | Date/ Day[1] | Time | Specimen<br>Type | Result |
|---|---|---|---|---|---|
| XXX-YYYY | Screening | yyyy-mm-dd/ xxx | hh:mm | Urine | Negative |

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

Source: list SAS datasets used to create table M:\ $402C409\production\programs\tlf\L16\_2-23.sas$ 

DateTime

#### Note to programmer:

Sort by date and time within subject.

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-40

Listing 16.2-24: Clinical Laboratory Tests-Hematology - All Subjects

| Subject | Parameter | Reference |
|---|---|---|
| D | (Units) | Range Visit Date / Day[1] Result Normal Range Indicator |
| XXX-YYYY | Hemoglobin (g/dL) | xxx - xxx Screening YYYY-MM-DD/-XX XXXXXXXXX Normal |
| | Hematocrit (%) | xxx - xxx Screening YYYY-MM-DD/-XX XXXXXXXX High |

Programming note: Order the lab parameters the same as shown in CRF. Any unscheduled lab results should be presented with scheduled data in date order. Number of decimal places for results should be as reported by the lab.

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-24.sas

DateTi

#### Same shell for:

Listing 16.2-25: Clinical Laboratory Tests-Chemistry - All Subjects

Listing 16.2-26: Clinical Laboratory Tests-Urinalysis - All Subjects

<sup>[1]</sup> Day = Visit date - first dose date +1 if Visit is on/after first dose; Otherwise Day=Visit date - first dose date.

| Pacira Pharmaceuticals, Inc. EXPAREL | | 402-C-409<br>Statistical Analysis Plan |
|---|---|---|
| Pacira Pharmaceuticals Listing 16.2-27: Unique Adverse Even | (Page X of Y)<br>ts Terms and Associated Coded Terms | Protocol: 402-C-409 |
| MedDRA Terms | | |
| SOC | | |
| Preferred Term | <pre>Verbatim(s)</pre> | |
| SOC1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| PT1.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| PT1.2 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| SOC2 | | |
| PT2.1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |
| | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | |

Coded using MedDRA

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16\_2-27.sas

DateTime

Note to programmer: Sort by SOC and preferred term in alphabetical order

Pacira Pharmaceuticals, Inc.

EXPAREL

Statistical Analysis Plan

Pacira Pharmaceuticals (Page X of Y) Protocol: 402-C-409 Listing 16.2-28: Unique Medication Terms and Associated Coded Terms Who Drug Dictionary Terms ACT1 ACT2 ACT3 ACT4 Preferred name Verbatim(s) ATC1 ATC1.2 PN1.2.1 PN1.2.2 ATC2 ATC2.2 ATC2.3 ATC2.4 PN2.2.3.4.1 

Coded using Who Drug Dictionary

Source: list SAS datasets used to create table M:\402C409\production\programs\tlf\L16 2-28.sas

DateTime

Note to programmer: Sort by ATC1, ATC2, ATC3, ATC4 and preferred name in alphabetical order